CLINICAL TRIAL: NCT00649428
Title: Safety and Efficacy Study of Isolagen TherapyTM in the Treatment of Nasolabial Fold Wrinkles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IT-R-005
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-02

CONDITIONS: Bilateral Nasolabial Fold Wrinkles
Keywords: Treatment of moderate to severe bilateral nasolabial fold wrinkles

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Biological: Autologous Human Fibroblast (azficel-T)
- Control (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Autologous Human Fibroblast (azficel-T) — 1. Collection of 3 mm post auricular skin punch biopsies.
  2. Three injection treatments administered 5 ± 1 weeks apart on each side of the face.
  Other Names: LAVIV
  Arms: Active
Biological: Placebo — 1. Collection of 3 mm post auricular skin punch biopsies.
  2. Three injection visits administered 5 ± 1 weeks apart on each side of the face.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the safety profile and the treatment effect of Isolagen TherapyTM compared with placebo when administered to bilateral nasolabial fold wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Level of severity of bilateral nasolabial fold wrinkles meeting severity criteria as per protocol
* Level of subject dissatisfaction with both nasolabial fold wrinkles as per protocol
* Ability to comply with the study requirements
* Negative pregnancy test (Females)
* Healthy post-auricular skin for biopsy

Exclusion Criteria:

* Excessive dermatochalasis of the treatment area
* Inability to lessen the nasolabial fold wrinkles by physically spreading the area apart
* Total area to be treated exceeds 20 cm in length
* Physical attributes which may prevent assessment or treatment as judged by the evaluator
* Use of an investigational product/procedure within 30 days prior to enrollment or plans for use during the study
* Previous treatment with the sponsor's product
* History of active autoimmune disease or organ transplantation
* Diagnosis of cancer, unless successfully treated or in remission (basal cell carcinoma is excluded)
* Active or chronic skin disease
* Known genetic disorders affecting fibroblasts or collagen
* Active systemic infection
* Requires chronic antibiotic or steroidal therapy
* Use of certain commercial products/procedures to the treatment area prior to study enrollment or plans for use during the study
* Use of systemic agents that increase bleeding or clotting, or disorders equated with these effects
* Known allergic reactions to agents used in preparation of treatment
* Excessive exposure to sun without adequate sun protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Total Skin & Beauty Dermatology Center, PC, Birmingham, Alabama
  - Silverburg Surgical & Medical Group, Newport Beach, California
  - Dermatology Research Institute, LLC, Coral Gables, Florida
  - River North Dermatology and Dermatologic Surgery, Naperville, Illinois
  - Aesthetic Solutions, Chapel Hill, North Carolina
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Center for Skin Research, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between October 23, 2006 and February 9, 2007.
Pre-assignment Details: Patients were enrolled and biopsied for manufacture of study product. All randomized patients were included in the Intent to Treat (ITT) population.
Groups:
- Autologous Fibroblasts: Patients treated with autologous dermal fibroblasts
- Placebo: Patients treated with placebo solution
Period: Overall Study
Arm/Group | Autologous Fibroblasts | Placebo
Started | 100 | 103
Completed | 80 | 88
Not Completed | 20 | 15
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 1 | 3
Not completed — Insufficient manufacturing yield | 5 | 1
Not completed — Protocol Violation | 6 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Fibroblasts | Placebo | Total
Number analyzed (Participants) | 100 | 103 | 203
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (8.32) | 55.9 (7.87) | 56.7 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 94 | 182
  Male | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 90 | 96 | 186
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 94 | 99 | 193
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 100 | 103 | 203

OUTCOME MEASURES:

1. Primary Outcome: Subject Wrinkle Assessment Responders
Description: A two point improvement on the Subject's live assessment of the wrinkles of the lower part of the face as compared to baseline on the Subject Wrinkle Assessment was considered a responder. The Subject Wrinkle Assessment scale was a five point scale with a score of -2 (Very Dissatisfied) being the worst and a score of +2 (Very Satisfied) being the best.
Time Frame: Baseline (prior to first treatment) and 6 months post final treatment
Population: Analysis population was the ITT population, defined as all randomized subjects.
Measure: Number; unit: participants
Groups:
- Autologous Fibroblast: Patients treated with autologous fibroblasts (azficel-T).
Arm/Group | Autologous Fibroblast | Placebo
Number analyzed (Participants) | 100 | 103
participants | 57 | 31
Statistical Analysis 1: Comparison: Autologous Fibroblast vs Placebo; A 5% level of significance was used as the threshold for determination of statistical significance, and all tests were two-tailed. the effect size and associated 95% confidence interval (CI) are provided for all comparative efficacy outcomes. Primary analysis of the two co-primary efficacy endpoints and the secondary efficacy endpoints were performed on the ITT population; Test type: Superiority or Other; p = .00001, Cochran-Mantel-Haenszel; Stratified by combined treatment site

2. Secondary Outcome: Subject Wrinkle Assessment Responders
Description: as for outcome 1
Time Frame: Baseline (prior to first treatment) compared to 3rd treatment visit, 2 and 4 months post final treatment
Population: Analysis population was the ITT population, defined as all randomized subjects.
Measure: Number; unit: participants
Groups:
- Autologous Fibroblasts: Patients treated with autologous fibroblasts (azficel-T).
Arm/Group | Autologous Fibroblasts | Placebo
Number analyzed (Participants) | 100 | 103
participants
  Responders at 3rd Treatment | 38 | 23
  Responders - 2 months Post Final Treatment | 49 | 25
  Responders - 4 months Post Final Treatment | 48 | 26

3. Secondary Outcome: Evaluator Wrinkle Severity Assessment Responders
Description: A responder was defined as a two point improvement on the blinded Evaluator's live assessment of each of the bilateral nasolabial fold wrinkles at rest using the 6-point ordinal Lemperle Wrinkle Severity Scale. On the Lemperle scale, a score of 5 (Very Deep Wrinkle) is worst and a score of 0 (No Visible Wrinkle) is best.
Time Frame: Baseline (prior to first treatment) compared to 3rd treatment visit, 2 and 4 months post final treatment
Population: Analysis population was the ITT population, defined as all randomized subjects.
Measure: Number; unit: participants
Arm/Group | Autologous Fibroblasts | Placebo
Number analyzed (Participants) | 100 | 103
participants
  Responders at 3rd Treatment | 14 | 5
  Responders - 2 months Post Final Treatment | 28 | 10
  Responders - 4 months Post Final Treatment | 27 | 9

4. Primary Outcome: Evaluator Wrinkle Severity Assessment Responders
Description: as for outcome 3
Time Frame: Baseline (prior to first treatment) and 6 months after last treatment
Population: Analysis population was the ITT population, defined as all randomized subjects.
Measure: Number; unit: participants
Arm/Group | Autologous Fibroblasts | Placebo
Number analyzed (Participants) | 100 | 103
participants | 33 | 7
Statistical Analysis 1: Comparison: Autologous Fibroblasts vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .00001, Cochran-Mantel-Haenszel; Stratified by combined treatment site

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the baseline visit through the final study visit, 6 months after final study treatment.
Arm/Group | Autologous Fibroblasts | Placebo
Serious Adverse Events (participants affected / at risk) | 2/100 | 4/103
Other Adverse Events (participants affected / at risk) | 32/100 | 34/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Fibroblasts (N=100) | Placebo (N=103)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adenocarcimona (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Athralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Chemical Abuser (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Fibroblasts (N=100) | Placebo (N=103)
Injection Site Bruising (General disorders) | 4 (5) | 12 (17)
Injection Site Erythema (General disorders) | 23 (53) | 17 (28)
Injection Site Pain (General disorders) | 5 (6) | 4 (5)
Injection Site Swelling (General disorders) | 18 (41) | 15 (27)
Nasopharyngitis (Infections and infestations) | 6 (6) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications or presentations by the Investigator or his associates, were required to be submitted to the sponsor for review and approval.